CLINICAL TRIAL: NCT01068197
Title: Low Glycemic Load Diets in Latino Children at Risk for Type 2 Diabetes
Acronym: COOL Kids
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nazrat Mirza (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH); Consumer Health Foundation (Unknown); Jessie Ball DuPont Foundation (Unknown)
Responsible Party: Sponsor-Investigator, Nazrat Mirza, Associate Professor, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K23RR022227; IRB # 3195; K23RR022227 (NIH)
Record Dates: First submitted 2010-02-11; First posted 2010-02-12 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Obesity; Type 2 Diabetes Mellitus
Keywords: Low Glycemic Load diet; Low Glycemic Index diet; Low Fat diet; Obese Hispanic American children and adolescents; At risk for type 2 diabetes mellitus
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low glycemic load dietary plan (Experimental): The subjects and their parents will be given instructions, and specific examples, to lower the glycemic load of their diets by replacing high-GI sources of carbohydrates with low-GI food sources, replacing energy from carbohydrate with energy from protein and fat, and attempt to balance meals and snacks with low-GI carbohydrate, proteins and low-fat food sources. The objective will be to achieve macronutrient composition for the low-GL diet of 45-50% low-GI carbohydrates, 20-25% protein, and 30-35% fat. All subjects will receive sessions on behavior modification, increasing physical activity and reducing sedentary behavior.
  At 3 months, subjects will be admitted to the GCRC for a 24 hour period for a meal study. They will be given standardized low-glycemic load diet for dinner, breakfast and lunch, followed by an ad lib snack platter. Their subjective, hormonal and metabolic responses will be serially measured.
  Interventions: Behavioral: Low Glycemic Load Diet versus Low Fat Diet
- Low fat diet (Active Comparator): For the low fat diet, subjects and their parents will be given instructions, and specific examples, to lower the fat content of their diet. The composition of the low-fat diet will be targeted to achieve 55-60% carbohydrates (with no discrimination by their glycemic index), 15-20% protein and 25-30% fat. All recruited children will receive sessions on behavior modification, increasing physical activity and reducing sedentary behavior.
  At 3 months, subjects will be admitted to the GCRC for a 24 hour period for a meal study. They will be given standardized high-glycemic load diet for dinner, breakfast and lunch, followed by an ad lib snack platter. Their subjective, hormonal and metabolic responses will be serially measured.
  Interventions: Behavioral: Low Glycemic Load Diet versus Low Fat Diet

INTERVENTIONS:
Behavioral: Low Glycemic Load Diet versus Low Fat Diet — We propose a randomized controlled clinical trial to evaluate the effectiveness of a low-glycemic load diet versus low-fat diet on insulin sensitivity, body composition, and other hormonal and biochemical measures. The culturally competent and family-based Intervention program has a dietary experimental component (low-glycemic load versus low-fat diet), as well as elements of physical activity, reduction in sedentary behavior and behavior modification. The nutrition training sessions are divided into 12 modules taught over a 12-week course. Care has been taken to make the content and intensity of the low-fat and low-glycemic load programs comparable. Both treatments include 12 weekly sessions, followed by nine monthly, and four 3-monthly sessions.
  Participants are obese (BMI ≥95th percentile for age and sex) Hispanic American children ages 7-14 years.

SUMMARY:
The purpose of this study are to:

1. compare two diet plans - a low-glycemic load (low-GL) diet and a low-fat diet. A low-GL diet is expected to keep blood sugar levels more normal, and because the sugar levels stay normal, prevent rapid rises of insulin in the blood. We want to test if Hispanic children at-risk for type 2 diabetes who are given a low-GL diet will have less insulin resistance, will lose more weight, and will decrease their chance of getting type 2 diabetes.
2. compare the effects of Low-GL and high-GL meals on appetitive, hormonal, and metabolic responses of obese Hispanic youth under controlled, standardized conditions. We want to test if children fed low-GL meals would have lower glucose and lower insulin responses, report less hunger and consume less energy than those fed high-GL meals.

DETAILED DESCRIPTION:
Overweight among minority children and adolescents is now the most prevalent pediatric public health problem in the United States. Our preliminary studies have found the prevalence of overweight among Hispanic children and adolescents in Washington DC is more than twice the U.S. national average. It is well established that overweight is associated with both medical and psychosocial complications, particularly for minority populations. Study of overweight Hispanic children has shown that they are at high risk for insulin resistance and impaired glucose tolerance (IGT), with IGT present in 28% of overweight Latino children with a family history of type 2 diabetes (T2DM). Despite the urgency to develop effective strategies to treat obesity and prevent T2DM in such children, few randomized controlled trials of weight management have been conducted in Hispanic children. Hence, there is an urgent need to develop effective, feasible and culturally competent obesity treatment programs targeted to Hispanic youth who are at great risk for obesity-associated co-morbidities, and who represent the fastest growing segment of the U.S. population.

A low-glycemic index (GI) or glycemic load (GL) diet is a much discussed, but quite controversial treatment of obesity. Some, but not all epidemiological studies show lower risk of diabetes among individuals consuming a low-GL diet. Short-term clinical studies examining the hormonal and biochemical responses to a low-GI diet have documented a reduction of reactive hyperglycemia and hyperinsulinemia, and decrease food intake. We propose that a low GL diet may be a particularly effective dietary regimen for overweight Latino children at risk for T2DM, who have a high consumption of processed and refined carbohydrate foods. The overall aim of this project is to determine the hormonal, metabolic, and body composition changes that occur during a two-year period of consumption of low-GL meals compared to low fat meals among Latino children at risk for T2DM. Our specific aims are:

- Specific Aim 1: To study the short- and long-term effects of a low-GL diet on insulin sensitivity in overweight Latino children at risk for T2DM.

Hypothesis 1: Insulin sensitivity will increase to a greater extent in children randomized to a low-GL diet than in children randomized to a reduced-fat meal prescription after 3, 12, and 24 months. The increase in insulin sensitivity found with a low-GL diet will not be fully explained by changes in BMI alone.

- Specific Aim 2: To determine the short- and long-term effects of a low-GL diet on BMI z-score and body fat changes in overweight Latino children at risk for T2DM.

Hypothesis 2: BMI z-score and body fat proportion will decrease to a greater extent in children randomized to a low-GL diet than in children randomized to a reduced-fat meal prescription after 3, 12, and 24 months observation periods.

- Specific Aim 3: To examine the effects of low-GL diet on markers of metabolic risk in overweight Latino children at risk for T2DM.

Hypothesis 3: Both traditional risk factors (e.g. systolic blood pressure, LDL-cholesterol, and triglycerides) and non-traditional risk factors (e.g. inflammatory [C-reactive protein, fibrinogen, and Plasminogen activating inhibitor -1], and adipocyte-derived factors [adiponectin, resistin, and free fatty acids]), related to insulin sensitivity will be lower in the low-GL meal group compared to the reduced-fat meal group at 3, 12, and 24 months.

- Specific Aim 4: To examine the subjective, hormonal, and metabolic responses of obese Hispanic youth to consumption of low-glycemic load and high glycemic load meals under controlled, standardized conditions.

Hypothesis 4: compared to the group fed high glycemic load meals, the low glycemic load group will have lower glucose and lower insulin responses, the low glycemic load group will report less hunger before their meals and greater satiety after their meals, and the low glycemic load group will consume less energy from a post-meal ad libitum snack platter.

Latino children ages 7-14y with BMI≥95th percentile and at-risk for T2DM will be randomly assigned either to a low-GL or a low-fat dietary plan for 2 years. Subjects will also participate in a culturally competent, family-based intervention program which includes behavior modification and enhanced physical activity. The frequence of intervention will consist of weekly visits for 12 weeks (Phase 1), monthly visits for 9 months (Phase 2), and 3-monthly visits for 12 months (Phase 3).

After completion of Phase 1, subjects will be admitted to the GCRC over a 24-hour period to participate in a meal study. Subjects will be provided with standardized meals consisting of either low-glycemic load (to the low-GL group) or high-glycemic load (to the high-GI group), and their subjective, hormonal, and metabolic responses will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Hispanic children aged 7-14 years with BMI >= 95th percentile at risk for T2DM and who are otherwise healthy
* Ethnicity will be by self-identification with the Hispanic or Latino cultural group by the subject's parents and both sets of grandparents.
* At risk for T2DM defined as a positive family history of T2DM plus insulin resistance (fasting hyperinsulinemia ≥ 15 uIU/mL) or impaired glucose tolerance (fasting glucose >110 mg/dl, or 2-hour postglucose challenge >140 mg/dl).
* Only one child per family will be eligible to participate in the study

Exclusion Criteria:

* pre-existing T2DM
* Cushing syndrome
* untreated hypothyroidism
* pervasive developmental disorder
* severe asthma
* severe untreated depression
* use of medications that promote weight gain or loss
* obesity-associated genetic syndromes (e.g. Prader Willi syndrome)

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 113 (Actual)
Dates: Start 2003-10; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Change in insulin sensitivity between the two dietary arms | at 3-, 12- and 24 months
Change in BMI z-score between the two dietary groups | 3-, 12-, and 24 months

SECONDARY OUTCOMES:
Change in body fat mass, lipid assay (LDL cholesterol, TG, FFA) between the two dietary arms | 3-, 12-, and 24 months
Differences in subjective, hormonal, and metabolic between the two dietary arms | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Nazrat M Mirza, MD, ScD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Mirza NM, Palmer MG, Sinclair KB, McCarter R, He J, Ebbeling CB, Ludwig DS, Yanovski JA. Effects of a low glycemic load or a low-fat dietary intervention on body weight in obese Hispanic American children and adolescents: a randomized controlled trial. Am J Clin Nutr. 2013 Feb;97(2):276-85. doi: 10.3945/ajcn.112.042630. Epub 2012 Dec 19. PMID 23255569
- [Derived] Mirza NM, Klein CJ, Palmer MG, McCarter R, He J, Ebbeling CB, Ludwig DS, Yanovski JA. Effects of high and low glycemic load meals on energy intake, satiety and hunger in obese Hispanic-American youth. Int J Pediatr Obes. 2011 Jun;6(2-2):e523-31. doi: 10.3109/17477166.2010.544740. Epub 2011 Feb 10. PMID 21309658